CLINICAL TRIAL: NCT02075255
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase 3 Efficacy and Safety Study of Benralizumab (MEDI-563) to Reduce Oral Corticosteroid Use in Patients With Uncontrolled Asthma on High Dose Inhaled Corticosteroid Plus Long-acting β2 Agonist and Chronic Oral Corticosteroid Therapy (ZONDA)
Brief Title: Efficacy and Safety Study of Benralizumab to Reduce OCS Use in Patients With Uncontrolled Asthma on High Dose Inhaled Corticosteroid Plus LABA and Chronic OCS Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00020
Record Dates: First submitted 2014-02-14; First posted 2014-03-03 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases, OCS, Oral Corticosteroids
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Benralizumab Arm A (Experimental): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab
- Benralizumab Arm B (Experimental): Benralizumab administered subcutaneously every 4 weeks for the first 3 dose and then every 8 weeks; matching placebo subcutaneously at the 4 week interim to maintain the blind.
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously every 4 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab administered subcutaneously every 4 weeks
  Arms: Benralizumab Arm A
Biological: Placebo — Placebo subcutaneously on study week 0 until study week 24 inclusive.
  Arms: Placebo
Biological: Benralizumab — Benralizumab administered subcutaneously every 4 weeks for the first 3 dose and then every 8 weeks; matching placebo subcutaneously at the 4 week interim to maintain the blind.
  Arms: Benralizumab Arm B

SUMMARY:
The purpose of this trial is to confirm if benralizumab can reduce the use of maintenance OCS in systemic corticosteroid dependent patients with severe refractory asthma with elevated eosinophils.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Female and male aged from 18 to 75 years, inclusively.
3. History of physician-diagnosed asthma requiring treatment with medium dose ICS and LABA.
4. Elevated level of peripheral blood eosinophil
5. Documented treatment with high-dose ICS and LABA for at least 6 months prior to Visit 1
6. Chronic oral corticosteroid therapy for at least 6 continuous months directly preceding Visit 1. Subjects must be on doses equivalent to 7.5 - 40 mg/day of prednisolone/prednisone at Visit 1 and be on a stable dose for at least 2 weeks prior to randomization. Patients must agree to switch to study required prednisone/prednisolone as their oral corticosteroid for the duration of the study.
7. Patients with documented failures of OCS reduction within 6 months prior to Visit 1 will not be required to proceed through the dose optimization phase during run-in.
8. Morning pre-bronchodilator (Pre-BD) FEV1 of <80% predicted
9. Evidence of asthma as documented by either:

   Airway reversibility (FEV1 ≥12% and 200 mL) demonstrated at Visit 1, Visit 2, or Visit 3 using the Maximum Post-bronchodilator Procedure OR Documented reversibility in the previous 24 months prior to Visit 1 OR Airway hyperresponsiveness (PC20 FEV1 methacholine concentration ≤8mg/mL) documented in the previous 12 months prior to planned date of randomization OR Airflow variability in clinic FEV1 ≥20% between 2 consecutive clinic visits documented in the 12 months prior to the planned date of randomization (FEV1 recorded during an exacerbation should not be considered for this criterion).

   All patients must have reversibility testing performed before randomization to establish a baseline characteristic.

   If patients do not demonstrate airway reversibility at either Visit 1 or Visit 2 and this is needed to qualify the patient for randomization, the site should reiterate the need to withhold short- and long-acting bronchodilators prior to Visit 3 in an effort to meet this inclusion criterion.
10. At least 1 documented asthma exacerbation in the previous 12 months prior to the date informed consent is obtained
11. Optimized OCS dose reached at least 2 weeks prior to randomization
12. Additional asthma controller medication must not have been initiated during run in/optimization period (not applicable for management of exacerbations during screening/ run in optimization phase)
13. At least 70% compliance with OCS use
14. At least 70% compliance with usual asthma controller ICS-LABA
15. Minimum 70% (i.e. 10 of 14 days) compliance with asthma daily diary (morning and evening diary)

Exclusion criteria:

1. Clinically important pulmonary disease other than asthma or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts.
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period
4. Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during run-in/optimization period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study
5. History of life-threatening asthma
6. Asthma control reached at an OCS dose of ≤5mg during run-in/OCS optimization phase
7. Qualifies for 3 consecutive dose reductions at Visits 2-4 and continues to meet OCS dose reduction criteria at Visit 5
8. Receipt of oral corticosteroids, other than prednisone or prednisolone, as the maintenance oral steroid controller for asthma symptoms from Visit 1 and throughout the study.
9. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.5 times the upper limit of normal (ULN) confirmed during screening period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD,PhD,FRCP,FRCPC, Principal Investigator — St Joseph's Healthcare Hamilton Firestone Institute for Respiratory Health 50 Charlton Avenue East Hamilton
Locations (77):
- United States (19):
  - Research Site, Los Angeles, California
  - Research Site, Centennial, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Iowa City, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Rochester, Minnesota
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Madison, Wisconsin
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Florida
  - Research Site, Mendoza
- Bulgaria (6):
  - Research Site, Kozloduy
  - Research Site, Pazardzhik
  - Research Site, Petrich
  - Research Site, Rousse
  - Research Site, Samokov
  - Research Site, Vratsa
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (6):
  - Research Site, Quillota
  - Research Site, Rancagua
  - Research Site, Santiago
  - Research Site, Talca
  - Research Site, Talcahuano
  - Research Site, Valparaíso
- France (6):
  - Research Site, Brest
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (7):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Großhansdorf
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Mainz
- Poland (10):
  - Research Site, Bydgoszcz
  - Research Site, Karczew
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Trzebnica
  - Research Site, Wroclaw
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (2):
  - Research Site, Málaga
  - Research Site, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
- Ukraine (5):
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Vinnytsia

REFERENCES:
- [Background] Nair P, Wenzel S, Rabe KF, Bourdin A, Lugogo NL, Kuna P, Barker P, Sproule S, Ponnarambil S, Goldman M; ZONDA Trial Investigators. Oral Glucocorticoid-Sparing Effect of Benralizumab in Severe Asthma. N Engl J Med. 2017 Jun 22;376(25):2448-2458. doi: 10.1056/NEJMoa1703501. Epub 2017 May 22. PMID 28530840
- [Derived] Menzies-Gow A, Hoyte FL, Price DB, Cohen D, Barker P, Kreindler J, Jison M, Brooks CL, Papeleu P, Katial R. Clinical Remission in Severe Asthma: A Pooled Post Hoc Analysis of the Patient Journey with Benralizumab. Adv Ther. 2022 May;39(5):2065-2084. doi: 10.1007/s12325-022-02098-1. Epub 2022 Mar 14. PMID 35287231
- [Derived] Menzies-Gow A, Corren J, Bel EH, Maspero J, Heaney LG, Gurnell M, Wessman P, Martin UJ, Siddiqui S, Garcia Gil E. Corticosteroid tapering with benralizumab treatment for eosinophilic asthma: PONENTE Trial. ERJ Open Res. 2019 Sep 25;5(3):00009-2019. doi: 10.1183/23120541.00009-2019. eCollection 2019 Jul. PMID 31579676
- [Derived] Chupp G, Lugogo NL, Kline JN, Ferguson GT, Hirsch I, Goldman M, Zangrilli JG, Trudo F. Rapid onset of effect of benralizumab on morning peak expiratory flow in severe, uncontrolled asthma. Ann Allergy Asthma Immunol. 2019 May;122(5):478-485. doi: 10.1016/j.anai.2019.02.016. Epub 2019 Feb 23. PMID 30802500
- See also: CSP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2559&filename=Nair_ZONDA_CSP_REDACTED.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 369 participants signed informed consent. 271 entered run in/OCS optimization period. 220 participants were randomized to receive treatment with benralizumab 30 mg Q4W, Q8W, or placebo. Of the 220 patients randomised, all (100.0%) received treatment with study drug
Groups:
- Benralizumab 30 mg q.4 Weeks: Benralizumab administered subcutaneously every 4 weeks
- Benralizumab 30 mg q.8 Weeks: Benralizumab administered subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks
- Placebo: Placebo administered subcutaneously
Period: Overall Study
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Started | 72 | 73 | 75
Completed | 68 | 69 | 72
Not Completed | 4 | 4 | 3
Not completed — Study specific withdrawal criteria | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo | Total
Number analyzed (Participants) | 72 | 73 | 75 | 220
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (12.0) | 52.9 (10.1) | 49.9 (11.7) | 51.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 48 | 135
  Male | 32 | 26 | 27 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage Reduction in Final OCS Dose Compared With Baseline While Maintaining Asthma Control
Description: Baseline OCS dose is the dose upon which the patient is stabilised at randomisation (Week 0). Final OCS dose is the dose at Week 28. The percentage reduction from baseline is defined as: {(Baseline dose-final dose)/baseline dose}*100%. If a patient discontinues from the study during a given dose reduction period, or the patient experiences an exacerbation between Weeks 24 and 28 or immediately before discontinuation, then the final OCS dose will be 1 dose level higher than that which directly preceded the event.
Time Frame: Week 28
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Percent
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Percent | 75.00 [50.00 to 83.30] | 75.00 [60.00 to 87.50] | 25.00 [0.00 to 33.30]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 33.3, 95% CI 2-sided [16.70 to 50.00] — Hodges-Lehmann estimate is used
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 37.50, 95% CI 2-sided [20.80 to 50.00] — Hodges Lehmann estimate is used

2. Secondary Outcome: Number and Percentage of Patients in Different Categories of Percent Reduction From Baseline in Final OCS Dose While Maintaining Asthma Control
Description: Number and percentage of patients in different categories of percent reduction from baseline in final OCS dose.
Time Frame: Week 28
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants
  >=90% reduction | 24 | 27 | 9
  >=75% reduction | 38 | 37 | 15
  >=50% reduction | 48 | 48 | 28
  >0% reduction | 55 | 58 | 40
  No change or any increase | 17 | 15 | 35
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, proportional odds model; Controlling for treatment group, region, and baseline OCS dose; Odds Ratio (OR) = 4.09, 95% CI 2-sided [2.22 to 7.57]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, proportional odds model; Controlling for treatment group, region, and baseline OCS dose; Odds Ratio (OR) = 4.12, 95% CI 2-sided [2.22 to 7.63]

3. Secondary Outcome: Percentage Reduction in Final OCS Dose Compared With Baseline While Maintaining Asthma Control for Patients With Baseline Eosinophils >=300/uL
Description: as for outcome 1
Time Frame: Week 28
Population: Full analysis set, baseline blood eosinophil >=300/uL
Measure: Median (95% Confidence Interval); unit: Percent
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 62 | 61 | 64
Percent | 75.00 [60.00 to 100.00] | 75.00 [60.00 to 91.70] | 0.00 [0.00 to 28.60]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 50.00, 95% CI 2-sided [25.00 to 66.70] — Hodges Lehmann estimate is used
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 50.00, 95% CI 2-sided [25.00 to 66.70] — Hodges Lehmann estimate is used

4. Secondary Outcome: The Percentage of Patients With ≥50% Reduction in Average Daily OCS Dose at Visit 14 Compared With Baseline Dose at Visit 6, While Maintaining Asthma Control
Description: as for outcome 1
Time Frame: Week 28
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants | 48 | 48 | 28
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 3.59, 95% CI 2-sided [1.79 to 7.22]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.57 to 5.86]

5. Secondary Outcome: The Proportion of Eligible Patients With ≥100% Reduction in Average Daily OCS Dose at Visit 14 Compared With Baseline Dose at Visit 6, While Maintaining Asthma Control
Description: as for outcome 1
Time Frame: Week 28
Population: Full analysis set, eligible for 100% reduction (ie, patients with baseline OCS dose <= 12.5 mg)
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 39 | 42 | 42
Participants | 22 | 22 | 8
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 5.23, 95% CI 2-sided [1.92 to 14.21]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 4.19, 95% CI 2-sided [1.58 to 11.12]

6. Secondary Outcome: The Proportion of Patients With ≤5.0 mg Reduction on Daily OCS Dose at Visit 14 Compared With Baseline Dose at Visit 6, While Maintaining Asthma Control.
Description: Baseline OCS dose is the dose upon which the patient is stabilised at randomisation (Week 0). Final OCS dose is the dose at Week 28. If a patient discontinues from the study during a given dose reduction period, or the patient experiences an exacerbation between Weeks 24 and 28 or immediately before discontinuation, then the final OCS dose will be 1 dose level higher than that which directly preceded the event.
Time Frame: Week 28
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants | 22 | 25 | 38
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.21 to 0.83]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.053, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.27 to 1.01]

7. Secondary Outcome: The Proportion of Patients With Average Final OCS Dose ≤5.0 mg Daily at Visit 14, While Maintaining Asthma Control
Description: Final OCS dose is the dose at Week 28. If a patient discontinues from the study during a given dose reduction period, or the patient experiences an exacerbation between Weeks 24 and 28 or immediately before discontinuation, then the final OCS dose will be 1 dose level higher than that which directly preceded the event.
Time Frame: Week 28
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants | 44 | 43 | 25
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 3.16, 95% CI 2-sided [1.60 to 6.23]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.41 to 5.31]

8. Secondary Outcome: Number and Percentage of Patients With ≥1 Asthma Exacerbation
Description: Number and percentage of patients with at least one post randomisation asthma exacerbation.
Time Frame: Immediately following the randomisation through Study Week 28
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants | 19 | 17 | 39
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.16 to 0.65]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for region; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.14 to 0.56]

9. Secondary Outcome: Time to the First Asthma Exacerbation
Description: Time to the first occurrence of asthma exacerbation post randomisation
Time Frame: The time from randomisation to the date of first asthma exacerbation over 28 weeks
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Days | NA [NA to NA] — median survival time is not estimable due to number of exacerbations had not reached 50%. | NA [NA to NA] — median survival time is not estimable due to number of exacerbations had not reached 50%. | 155 [111 to NA] — Upper 95% CI for median is not estimable due to the curve representing the upper confidence limit of the survival function is above 50%
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Cox; Including covariates treatment group, region, number of exacerbations in the previous year; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.22 to 0.66]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Cox; Including covariates treatment group, region, number of exacerbations in the previous year; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.17 to 0.57]

10. Secondary Outcome: Time to the First Asthma Exacerbation Requiring Hospitalization or ER Visit
Description: Time to the first exacerbation requiring hospitalization or ER visit post randomisation
Time Frame: The time from randomisation to the date of first asthma exacerbation associated with hospitalization or ER over 28 weeks.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Days | NA [NA to NA] — median survival time is not estimable due to number of exacerbations resulting hospitalization or ER visit had not reached 50%. | NA [NA to NA] — median survival time is not estimable due to number of exacerbations resulting hospitalization or ER visit had not reached 50%. | NA [NA to NA] — median survival time is not estimable due to number of exacerbations resulting hospitalization or ER visit had not reached 50%.
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.291, Regression, Cox; Including covariates treatment group, region, any exacerbations in the previous year requiring hospitalization or ER visit; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.14 to 1.64]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.042, Regression, Cox; [statistical method as in outcome 10, analysis 1]; Hazard Ratio (HR) = 0.12, 95% CI 2-sided [0.01 to 0.63]

11. Secondary Outcome: The Annualized Rate of Asthma Exacerbation
Description: The annualized exacerbation rate is based on unadjudicated exacerbation reported by the investigator adjusted by the time of follow-up.
Time Frame: The time from randomisation to the date of week 28 visit (end of treatment) or last contact if the patient is lost to follow up
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
events/year | 0.83 [0.55 to 1.26] | 0.54 [0.34 to 0.88] | 1.83 [1.33 to 2.50]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.003, negative binomial model; Including covariates treatment group, region, number of exacerbations in the previous year. The log of follow-up time is used as offset variable; Rate ratio = 0.45, 95% CI 2-sided [0.27 to 0.76]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, negative binomial model; [statistical method as in outcome 11, analysis 1]; Rate ratio = 0.3, 95% CI 2-sided [0.17 to 0.53]

12. Secondary Outcome: The Annualized Rate of Asthma Exacerbations That Are Associated With an Emergency Room Visit or a Hospitalization
Description: The annualized exacerbation rate is based on unadjudicated exacerbation reported by the investigator that are associated with an emergency room visit or a hospitalization adjusted by the time of follow-up.
Time Frame: as for outcome 11
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
events/year | 0.14 [0.05 to 0.38] | 0.02 [0.00 to 0.18] | 0.32 [0.16 to 0.65]
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.187, negative binomial model; Covariates include treatment, region, any exacerbations in the previous year requiring hospitalization/ER. Log of follow-up time is the offset; Rate ratio = 0.44, 95% CI 2-sided [0.13 to 1.49]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.018, negative binomial model; [statistical method as in outcome 12, analysis 1]; Rate ratio = 0.07, 95% CI 2-sided [0.01 to 0.63]

13. Secondary Outcome: Number of Days in Hospital Due to Asthma
Description: Number of days in hospital due to asthma, if none, 0 day is considered
Time Frame: as for outcome 11
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Days | 0.3 (1.41) [0.02 to 0.19] | 0.5 (3.86) [0.00 to 0.08] | 1.2 (6.66) [0.04 to 0.35]

14. Secondary Outcome: Change From Baseline to Week 28 in Pre-bronchodilator FEV1
Description: Baseline is defined as the last non-missing value prior to the first dose of study treatment. Change from baseline to Week 28 in two treatment groups is compared to placebo group.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 68 | 68 | 73
Liter | 0.230 (0.429) | 0.255 (0.508) | 0.114 (0.401)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.153, Mixed Models Analysis; Including covariates: treatment group, region, baseline pre-BD FEV1 value, visit, and visit by treatment interaction; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [-0.040 to 0.251]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.129, Mixed Models Analysis; Including covariates: treatment group, region, baseline pre-BD FEV1 value, visit, and visit by treatment interaction; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [-0.033 to 0.258]

15. Secondary Outcome: Change From Baseline to Week 28 in Asthma Symptom Scores (Total)
Description: Asthma symptoms during night time and daytime are recorded by the patient in the asthma daily diary. Symptom score values are from 0 (No asthma symptom) to 3 (unable to sleep because of asthma, or unable to do normal activities due to asthma), and total asthma symptom score is the sum of the daytime and night time score (0 to 6). Lower score (0) is indicating better asthma symptom, while higher score (6) is indicating worse asthma symptom. Baseline is defined as the average of data collected from the evening of study day -14 to the morning of study day 1. Each time point is calculated as bi-weekly means based on daily diary data. If more than 50% of scores are missing in a 14 day period then this is considered as missing. Symptom score lower is better.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 68 | 67
Scores on a scale | -0.58 (1.03) | -0.77 (1.03) | -0.58 (1.03)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.947, Mixed Models Analysis; Include covariates: treatment group, baseline asthma symptom score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.35 to 0.32]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.291, Mixed Models Analysis; Include covariates: treatment group, baseline asthma symptom score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.51 to 0.16]

16. Secondary Outcome: Change From Baseline to Week 28 in Asthma Symptom Scores (Daytime)
Description: Asthma symptoms during daytime are recorded by the patient in the asthma daily diary. Symptom score values are from 0 (No asthma symptom) to 3 (unable to sleep because of asthma, or unable to do normal activities due to asthma). Lower score (0) is indicating better asthma symptom, while higher score (3) is indicating worse asthma symptom. Baseline is defined as the average of data collected from the evening of study day -14 to the morning of study day 1. Each time point is calculated as bi-weekly means based on daily diary data. If more than 50% of scores are missing in a 14 day period then this is considered as missing. Symptom score lower is better.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 69 | 69
Scores on a scale | -0.32 (0.56) | -0.44 (0.52) | -0.32 (0.57)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.998, Mixed Models Analysis; Include covariates: treatment group, baseline asthma symptom score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.18 to 0.18]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.177, Mixed Models Analysis; Include covariates: treatment group, baseline asthma symptom score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.30 to 0.05]

17. Secondary Outcome: Change From Baseline to Week 28 in Asthma Symptom Scores (Nighttime)
Description: Asthma symptoms during night time are recorded by the patient in the asthma daily diary. Symptom score values are from 0 (No asthma symptom) to 3 (unable to sleep because of asthma, or unable to do normal activities due to asthma). Lower score (0) is indicating better asthma symptom, while higher score (3) is indicating worse asthma symptom. Baseline is defined as the average of data collected from the evening of study day -14 to the morning of study day 1. Each time point is calculated as bi-weekly means based on daily diary data. If more than 50% of scores are missing in a 14 day period then this is considered as missing. Symptom score lower is better.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 68 | 67
Scores on a scale | -0.27 (0.51) | -0.34 (0.54) | -0.27 (0.54)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.973, Mixed Models Analysis; Include covariates: treatment group, baseline asthma symptom score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.17 to 0.17]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.480, Mixed Models Analysis; Include covariates: treatment group, baseline asthma symptom score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.23 to 0.11]

18. Secondary Outcome: Change From Baseline to Week 28 in Rescue Medication Use
Description: Baseline is defined as the average of data collected from the evening of study day -14 to the morning of study day 1. Each timepoint is calculated as bi-weekly means based on daily diary data. If more than 50% of scores are missing in a 14 day period then this will be considered as missing. The number of inhalations (puffs) per day will be calculated as follows: Number of night inhaler puffs + 2 x [number of night nebulizer times] + number of day inhaler puffs + 2 x [number of day nebulizer times].
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: number of puffs per day
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 68 | 67
number of puffs per day | -1.39 (2.86) | -2.58 (4.36) | -1.07 (2.86)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.397, Mixed Models Analysis; Include covariates: treatment group, baseline total asthma rescue medication use, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.44 to 0.57]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; [statistical method as in outcome 18, analysis 1]; Mean Difference (Final Values) = -1.41, 95% CI 2-sided [-2.42 to -0.41]

19. Secondary Outcome: Change From Baseline to Week 28 in Home Lung Function (Morning Peak Expiratory Flow)
Description: Morning peak expiratory flow change from baseline to week 28. Baseline is defined as the average of data collected from the evening of study day -14 to the morning of study day 1. Each timepoint is calculated as bi-weekly means based on daily diary data.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Liter/min
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 68 | 67
Liter/min | 32.697 (89.457) | 43.022 (73.303) | 10.884 (69.356)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.143, Mixed Models Analysis; Include covariates: treatment group, baseline morning PEF, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = 19.25, 95% CI 2-sided [-6.58 to 45.07]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; Include covariates: treatment group, baseline morning PEF, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = 30.01, 95% CI 2-sided [4.26 to 55.76]

20. Secondary Outcome: Change From Baseline to Week 28 in Home Lung Function (Evening Peak Expiratory Flow)
Description: Evening peak expiratory flow change from baseline to week 28. Baseline is defined as the average of data collected from the evening of study day -14 to the morning of study day 1. Each timepoint is calculated as bi-weekly means based on daily diary data
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Liter/min
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 69 | 66
Liter/min | 21.885 (83.136) | 34.157 (69.287) | 2.933 (72.302)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.237, Mixed Models Analysis; Include covariates: treatment group, baseline evening PEF, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = 15.19, 95% CI 2-sided [-10.08 to 40.46]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; Include covariates: treatment group, baseline evening PEF, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = 31.52, 95% CI 2-sided [6.32 to 56.71]

21. Secondary Outcome: Change From Baseline to Week 28 in the Proportion of Nights With Awakening Due to Asthma Requiring Rescue Medication
Description: Baseline is defined as the proportion of nights from the evening of study day -14 to the morning of study day 1.Each timepoint is calculated as bi-weekly proportions based on daily diary data. If more than 50% of data are missing in a 14 day period then this will be considered as missing.Proportion of nights with noctural awakenings is defined as the number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with data.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Proportion
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 67 | 68 | 67
Proportion | -0.158 (0.283) | -0.2 (0.337) | -0.186 (0.344)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.742, Mixed Models Analysis; Including covariates: treatment group, baseline proportion of nights with noctural awakenings, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.08 to 0.11]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.693, Mixed Models Analysis; [statistical method as in outcome 21, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.11 to 0.07]

22. Secondary Outcome: Change From Baseline to Week 28 in ACQ-6
Description: ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses. Mean scores of <=0.75 indicates well-controlled asthma, scores between 0.75 to <=1.5 indicate partly controlled asthma, and >1.5 indicates not well controlled asthma.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 66 | 66 | 67
Scores on a scale | -0.86 (0.95) | -1.09 (1.09) | -0.68 (1.10)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.139, Mixed Models Analysis; Include covariates: treatment group, baseline ACQ-6 score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.55 to 0.08]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Include covariates: treatment group, baseline ACQ-6 score, region, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.86 to -0.23]

23. Secondary Outcome: ACQ-6 Responders (Improvement) at Week 28
Description: Improvement is defined as ACQ-6 (End of treatment - baseline) <= -0.5. No change is defined as ACQ-6 (End of treatment - baseline) >-0.5 and <0.5. Deterioration is defined as ACQ-6 (End of treatment - baseline) >= 0.5. ACQ-6 score is defined as the average of the first 6 items of the ACQ questionnaire on symptoms, activity limitations and rescue medication.Scores range from 0 (totally controlled) to 6 (severely uncontrolled). Baseline is defined as the last non-missing value prior to randomisation. End of treatment is defined as week 28. Patients with missing or non-evaluable ACQ-6 at week 28 are considered non-responder.
Time Frame: Week 28
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants | 41 (0.95) | 46 (1.09) | 41 (1.10)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.658, Regression, Logistic; Including covariates: treatment group, baseline ACQ-6 score, region, number of exacerbations in the previous year; Odds Ratio (OR) = 1.165, 95% CI 2-sided [0.592 to 2.295]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.155, Regression, Logistic; Including covariates: treatment group, baseline ACQ-6 score, region, number of exacerbations in the previous year; Odds Ratio (OR) = 1.661, 95% CI 2-sided [0.826 to 3.340]

24. Secondary Outcome: Change From Baseline at Week 28 in AQLQ(S)+12 (Overall)
Description: AQLQ(S)+12 overall score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. AQLQ(S)+12 is a 7-point scale questionnaire, ranging from 7 (no impairment) to 1 (severe impairment). Total or domain score change of >=0.5 are considered clinically meaningful.
Time Frame: Change from baseline at week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 66 | 67 | 68
Scores on a scale | 0.90 (0.93) | 1.05 (1.04) | 0.67 (1.10)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.151, Mixed Models Analysis; Including covariates: treatment group, region, baseline AQLQ(S)+12 score, visit, and treatment by visit interaction; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.08 to 0.53]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Including covariates: treatment group, region, baseline AQLQ(S)+12 score, visit, and treatment by visit interaction; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.14 to 0.76]

25. Secondary Outcome: AQLQ(s)+12 Responders (Improvement) at Week 28
Description: AQLQ(S)+12 overall score is defined as the average of all 32 questions in the AQLQ(S)+12 questionnaire. Improvement is defined as AQLQ(S)+12 (End of treatment - baseline)>=0.5. No change is defined as AQLQ(S)+12 (End of treatment - baseline) >-0.5 and <0.5. Deterioration is defined as AQLQ(S)+12 (End of treatment - baseline) <= -0.5. Baseline is defined as the last AQLQ(S)+12 score prior to randomisation. End of treatment is defined as week 28. Patients with missing or non-evaluable score at week 28 are considered as non-responder.
Time Frame: Week 28
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants | 43 (0.95) | 44 (1.09) | 39 (1.10)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p = 0.220, Regression, Logistic; Including covariates: treatment group, region, baseline AQLQ(S)+12 score, number of exacerbations in the previous year; Odds Ratio (OR) = 1.538, 95% CI 2-sided [0.773 to 3.060]
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p = 0.108, Regression, Logistic; Including covariates: treatment group, region, baseline AQLQ(S)+12 score, number of exacerbations in the previous year; Odds Ratio (OR) = 1.783, 95% CI 2-sided [0.882 to 3.605]

26. Secondary Outcome: Extent of Exposure
Description: Duration of exposure from first dose date to last dose date.
Time Frame: From first dose to Week 24
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Days | 162.53 (30.09) | 159.77 (35.781) | 167.05 (10.697)

27. Secondary Outcome: Serum Concentration of Benralizumab
Description: Pre-dose serum concentrations at each visit
Time Frame: Pre-first dose to Week 36
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 71 | 72 | 0
ng/mL
  Baseline (n=69, 71) | NA (NA) — Value is less than lower limit of quantification | NA (NA) — Value is less than lower limit of quantification |
  Week 4 (n=67, 71) | 804.37 (52.77) | 721.42 (52.30) |
  week 8 (n=66, 69) | 1152.96 (53.16) | 1019.65 (89.51) |
  Week 12 (n=68, 67) | 1319.14 (66.05) | 1057.91 (125.74) |
  Week 16 (n=67,67) | 1337.98 (118.90) | 303.54 (144.53) |
  Week 24 (n=65, 66) | 1162.62 (151.35) | 185.17 (278.32) |
  Week 28 (n=65, 65) | 1125.96 (173.79) | 684.57 (205.67) |
  Week 36 (n=2, 4) | 11.11 (2140.87) | 5.92 (1230.68) |

28. Secondary Outcome: Anti-drug Antibody Response
Description: Number and percentage of patients in different ADA response categories
Time Frame: From baseline to follow-up Week 36
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 72 | 73 | 75
Participants
  Positive at any visit | 5 | 7 | 6
  Baseline and Post-baseline Postive: number analyzed (Participants) | 68 | 69 | 75
  Baseline and Post-baseline Postive | 0 | 0 | 3
  Only post-baseline positive: number analyzed (Participants) | 71 | 70 | 75
  Only post-baseline positive | 5 | 6 | 3
  Only baseline positive: number analyzed (Participants) | 69 | 72 | 75
  Only baseline positive | 0 | 1 | 0
  Persistently positive: number analyzed (Participants) | 71 | 70 | 75
  Persistently positive | 4 | 6 | 5
  Transient positive: number analyzed (Participants) | 71 | 70 | 75
  Transient positive | 1 | 0 | 1

29. Secondary Outcome: Percent Change From Baseline in Blood Eosinophil Counts
Description: Percent change from baseline in blood eosinophil counts at week 28
Time Frame: Change from baseline at Week 28
Population: Full analysis set. Number of participants analyzed contains number of participants who had value at Week 28.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 63 | 62 | 66
percent change | -97.4 (12.93) | -94.9 (16.54) | 45.5 (239.51)
Statistical Analysis 1: Comparison: Benralizumab 30 mg q.4 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Include covariates: treatment group, baseline eosinophil count, region, visit, treatment by visit; Mean Difference (Final Values) = -162.2, 95% CI 2-sided [-220.1 to -104.3] — Percent change
Statistical Analysis 2: Comparison: Benralizumab 30 mg q.8 Weeks vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Include covariates: treatment group, baseline eosinophil count, region, visit, treatment by visit; Mean Difference (Final Values) = -159.4, 95% CI 2-sided [-217.9 to -100.9] — Percent change

30. Secondary Outcome: Total Lung Capacity
Description: Change from baseline in total lung capacity
Time Frame: From baseline to Week 28
Population: Global Sputum Substudy
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 22 | 26 | 23
Liter
  Week 12 (n=17, 23, 17) | -0.02 (0.95) | -0.07 (0.68) | -0.30 (1.08)
  Week 28 (n=14, 18, 15) | 0.11 (1.31) | -0.21 (0.70) | -0.47 (1.47)

31. Secondary Outcome: Residual Volume
Description: Change from baseline in residual volume
Time Frame: From baseline to Week 28
Population: Global Sputum Substudy
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 22 | 26 | 23
Liter
  Week 12 (n=17, 23, 17) | 0.02 (1.00) | -0.22 (0.74) | -0.35 (1.03)
  Week 28 (n=14, 18, 15) | 0.07 (1.34) | -0.31 (0.71) | -0.41 (1.27)

32. Secondary Outcome: Vital Capacity
Description: Change from baseline in vital capacity
Time Frame: From baseline to Week 28
Population: Global Sputum Substudy
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 22 | 26 | 23
Liter
  Week 12 (n=17, 24, 18) | 0.15 (0.80) | 0.18 (0.35) | 0.13 (0.89)
  Week 28 (n=14, 18, 15) | 0.15 (0.41) | 0.11 (0.48) | -0.08 (0.41)

33. Secondary Outcome: Functional Residual Capacity
Description: Change from baseline in functional residual capacity
Time Frame: From baseline to Week 28
Population: Global Sputum Substudy
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 22 | 26 | 23
Liter
  Week 12 (n=17,23, 18) | -0.05 (1.06) | -0.09 (0.74) | -0.38 (0.99)
  Week 28 (n=13,18, 15) | -0.15 (1.49) | -0.26 (0.74) | -0.43 (1.25)

34. Secondary Outcome: Inspiratory Capacity
Description: Change from baseline in inspiratory capacity
Time Frame: From baseline to Week 28
Population: Global Sputum Substudy
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg q.4 Weeks | Benralizumab 30 mg q.8 Weeks | Placebo
Number analyzed (Participants) | 22 | 26 | 23
Liter
  Week 12 (n=17, 23, 17) | 0.44 (1.22) | 0.14 (0.88) | -0.01 (0.40)
  Week 28 (n=14, 17, 15) | 0.52 (1.16) | 0.09 (1.01) | -0.02 (0.40)

ADVERSE EVENTS:
Time Frame: Include events occurred from the start of study treatment to the end of study (up to 36 weeks)
Groups:
- Benra 30 mg q.4 Weeks: Benralizumab administered subcutaneously every 4 weeks
- Benra 30 mg q.8 Weeks: Benralizumab administered subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Placebo
Serious Adverse Events (participants affected / at risk) | 7/72 | 7/73 | 14/75
Other Adverse Events (participants affected / at risk) | 34/72 | 34/73 | 49/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg q.4 Weeks (N=72) | Benra 30 mg q.8 Weeks (N=73) | Placebo (N=75)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg q.4 Weeks (N=72) | Benra 30 mg q.8 Weeks (N=73) | Placebo (N=75)
Vertigo (Ear and labyrinth disorders) | 1 (5) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 5 (7) | 8 (10) | 12 (13)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 11 (13) | 12 (14) | 15 (17)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Rhinitis (Infections and infestations) | 2 (2) | 6 (7) | 2 (2)
Sinusitis (Infections and infestations) | 5 (8) | 4 (5) | 8 (11)
Upper respiratory tract infection (Infections and infestations) | 4 (7) | 5 (6) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (5)
Headache (Nervous system disorders) | 5 (7) | 6 (10) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 1 (2) | 14 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.